CLINICAL TRIAL: NCT04661202
Title: Effects of Exercise Training on Pelvic Floor Symptoms and Function in Adults With Constipation: A Randomized Controlled Trial
Brief Title: Effects of Exercise Training on Pelvic Floor Symptoms and Function in Adults With Constipation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng Kung University (Other)
Responsible Party: Principal Investigator, Kuan-Yin Lin, Assistant professor, National Cheng Kung University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B-BR-109-090
Record Dates: First submitted 2020-12-03; First posted 2020-12-10 (Actual); Results first posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-02

CONDITIONS: Constipation
Keywords: constipation; resistance exercise; aerobic exercise; pelvic floor muscle training
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise training group (Experimental): * Aerobic exercise
  * Resistance exercise (including pelvic floor muscle training with biofeedback)
  * Stretching exercise
  * Home exercise
  Interventions: Other: multimodal exercise training
- Control group (No Intervention): ・Usual care
  After baseline assessment, the participants will receive health and lifestyle advices related to bowel symptoms, which include maintaining moderate physical activity, healthy diet, and ideal defecation posture, and establishing a personal bowel schedule and other behavioral changes that promote regular bowel movements.
  Upon request, the participants will be provided with the same intervention program as the exercise training group after 8 weeks participation.

INTERVENTIONS:
Other: multimodal exercise training — A supervised moderate-intensity exercise training session, which will include aerobic exercise with a stationary exercise bike, resistance exercise using dumbbell, theraband band, or gym ball for each major muscle groups and core muscles (including pelvic floor muscle (PFM) training with biofeedback), and stretching exercise, twice a week for 8 weeks. All exercises will be individualized based on participant's heart rate reserve and Rate of Perceived Exertion (RPE). An oximeter and a sphygmomanometer will be used to monitor the heart rate, oxygen saturation and blood pressure of the participants to ensure safety.
  A home exercise program will include a walking exercise for 30 minutes per day and a PFM training with the aim of completing 1~3 sets of 8~12 submaximal contraction of PFM by holding 6~10 seconds with 12~20 seconds of rest between each contraction, and it will end with 3 maximal PFM contractions by holding 1~3 seconds 3~6 seconds of rest between each contraction.
  Arms: Exercise training group

SUMMARY:
Constipation is a common problem in the general population. Defecation disorders caused by abnormal contraction or insufficient relaxation of the pelvic floor muscles during defecation may be one of the most possible causes of constipation. Although constipation is not life-threatening, it may have a significant impact on the quality of life. Aerobic exercise has been shown to improve symptoms of constipation in adults with constipation. However, there is no research investigating the effects of a multimodal exercise training on pelvic floor symptoms and pelvic floor muscle function in this population and only few studies have evaluated the pelvic floor muscle function using objective assessment tools among this population. The aim of the study is to investigate the effect of a multimodal exercise training program on constipation symptoms and pelvic floor muscle function in adults with constipation. The investigator will conduct a randomized controlled trial to evaluate the effectiveness of exercise training for adults with constipation. This study hypothesizes that (1) a multimodal exercise training can improve pelvic floor symptoms and function in adults with constipation, and (2) the improvement in exercise training group will be higher than that in control group.

DETAILED DESCRIPTION:
This is a randomized controlled trial. Adults with constipation will be recruited and randomly assigned to either the intervention group or the control group. The intervention group will receive 16 sessions of therapist-supervised, combined resistance (including pelvic floor muscle training) and aerobic exercise training twice weekly for 8 weeks. The control group will receive usual care. All participants will be assessed at baseline and post-intervention. The primary outcome measure is the severity of the patient's self-reported constipation symptoms measured using the Patient Assessment of Constipation Symptoms Questionnaire (PACSYM). The secondary outcomes are pelvic floor muscle function assessed through the Pelvic Floor Muscle Coordination Scale (PFMCS), digital rectal examination, and anorectal manometry; quality of life measured by the Patient Assessment of Constipation Quality of Life Questionnaire (PACQOL); and physical activity levels measured using the International Physical Activity Questionnaire (IPAQ). Intention-to-treat analysis will be performed to preserve the sample size and original randomization. Mann-Whitneyand Chi-square testsest will be used for continuota and categorical data to compare the baseline characteristics between the two groups. Wilcoxon signed-rank test and the Mann-Whitney U test will be used for intragroup and intergroup comparison of outcome variables. The p-value of < 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 20 years and 64 years
* Participants who fulfill the Rome IV criteria for constipation which include two or more of the following: a) straining > 25% of defecations; b) lumpy or hard stools > 25% of defecations; c) sensation of incomplete evacuation > 25% of defecations; d) sensation of anorectal obstruction/blockage > 25% of defecations; e) manual maneuvers to facilitate > 25% of defecations; f) < 3 spontaneous bowel movements per week
* Participants who have sufficient language skills to participate

Exclusion Criteria:

* Participants who have received exercise or pelvic floor muscle training under supervision in the past 12 months
* Participants with previous abdominal surgery, anorectal trauma or surgery, or previous diagnosis of neuropathy or anal sphincter dysfunction
* Presence of malignancies, severe cardiovascular disease or other severe physical/psychiatric impairments that prevent participation in the study
* Pregnant or within 12 months postpartum

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-03-23 (Actual); Study Completion 2022-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kuan-Yin Lin, PhD, Principal Investigator — National Cheng Kung University
Locations (1):
- National Cheng Kung University, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rao SS, Bharucha AE, Chiarioni G, Felt-Bersma R, Knowles C, Malcolm A, Wald A. Functional Anorectal Disorders. Gastroenterology. 2016 Mar 25:S0016-5085(16)00175-X 10.1053/j.gastro.2016.02.009. doi: 10.1053/j.gastro.2016.02.009. Online ahead of print. PMID 27144630
- [Background] Gao R, Tao Y, Zhou C, Li J, Wang X, Chen L, Li F, Guo L. Exercise therapy in patients with constipation: a systematic review and meta-analysis of randomized controlled trials. Scand J Gastroenterol. 2019 Feb;54(2):169-177. doi: 10.1080/00365521.2019.1568544. Epub 2019 Mar 7. PMID 30843436
- [Background] Virtuoso JF, Menezes EC, Mazo GZ. Effect of Weight Training with Pelvic Floor Muscle Training in Elderly Women with Urinary Incontinence. Res Q Exerc Sport. 2019 Jun;90(2):141-150. doi: 10.1080/02701367.2019.1571674. Epub 2019 Apr 4. PMID 30945991
- [Background] Frank L, Kleinman L, Farup C, Taylor L, Miner P Jr. Psychometric validation of a constipation symptom assessment questionnaire. Scand J Gastroenterol. 1999 Sep;34(9):870-7. doi: 10.1080/003655299750025327. PMID 10522604
- [Background] Sadowy AM, Brouwer HL, Finseth DL, Hagener KM, Lawrence AE, Hollman JH. Development of a Pelvic Floor Muscle Coordination Scale. Journal of Women's Health Physical Therapy. 2010;34(3):81-8.
- [Background] Gosling J, Plumb A, Taylor SA, Cohen R, Emmanuel AV. High-resolution anal manometry: Repeatability, validation, and comparison with conventional manometry. Neurogastroenterol Motil. 2019 Jun;31(6):e13591. doi: 10.1111/nmo.13591. PMID 31094054
- [Background] Kaushal JN, Goldner F. Validation of the digital rectal examination as an estimate of anal sphincter squeeze pressure. Am J Gastroenterol. 1991 Jul;86(7):886-7. PMID 2058632
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Marquis P, De La Loge C, Dubois D, McDermott A, Chassany O. Development and validation of the Patient Assessment of Constipation Quality of Life questionnaire. Scand J Gastroenterol. 2005 May;40(5):540-51. doi: 10.1080/00365520510012208. PMID 16036506

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the outpatient department of Colorectal Surgery of National Cheng Kung University Hospital, Tainan, Taiwan, the clinic, community, and social media from January 2021 to June 2022.
Groups:
- Exercise Training Group: * Aerobic exercise
  * Resistance exercise (including pelvic floor muscle training with biofeedback)
  * Stretching exercise
  * Home exercise
  Multimodal exercise training:
  A supervised moderate-intensity exercise training session, which will include aerobic exercise with a stationary exercise bike, resistance exercise using dumbbell, theraband band, or gym ball for each major muscle groups and core muscles (including pelvic floor muscle (PFM) training with biofeedback), and stretching exercise, twice a week for 8 weeks. All exercises will be individualized based on participant's heart rate reserve and Rate of Perceived Exertion (RPE). An oximeter and a sphygmomanometer will be used to monitor the heart rate, oxygen saturation and blood pressure of the participants to ensure safety.
  A home exercise program will include a walking exercise for 30 minutes per day and a PFM training with the aim of completing 1~3 sets of 8~12 submaximal contraction of PFM by holding 6~10 seconds with 12~20 seconds of rest between each contraction, and it will end with 3 maximal PFM contractions by holding 1~3 seconds 3~6 seconds of rest between each contraction.
- Control Group: ．Usual care
  After baseline assessment, the participants will receive health and lifestyle advices related to bowel symptoms, which include maintaining moderate physical activity, healthy diet, and ideal defecation posture, and establishing a personal bowel schedule and other behavioral changes that promote regular bowel movements.
  Upon request, the participants will be provided with the same intervention program as the exercise training group after 8 weeks participation.
Period: Overall Study
Arm/Group | Exercise Training Group | Control Group
Started | 14 | 13
Completed | 11 | 12
Not Completed | 3 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lack of Efficacy | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Control Group: ●Usual care
  After baseline assessment, the participants will receive health and lifestyle advices related to bowel symptoms, which include maintaining moderate physical activity, healthy diet, and ideal defecation posture, and establishing a personal bowel schedule and other behavioral changes that promote regular bowel movements.
  Upon request, the participants will be provided with the same intervention program as the exercise training group after 8 weeks participation.
- Total: Total of all reporting groups
Arm/Group | Exercise Training Group | Control Group | Total
Number analyzed (Participants) | 14 | 13 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.07 (12.47) | 37.92 (16.19) | 36.96 (14.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 11 | 24
  Male | 1 | 2 | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Height [Mean (Standard Deviation); unit: centimeter] | 161.6 (7.51) | 159.7 (6.12) | 160.7 (6.81)
Weight [Mean (Standard Deviation); unit: kilogram] | 59.5 (8.02) | 60.5 (16.66) | 60.0 (12.67)
Body mass index (BMI) [Mean (Standard Deviation); unit: kilogram/meter^2] | 22.8 (2.82) | 23.6 (5.43) | 23.2 (4.21)
Smoking status [Count of Participants; unit: Participants]
  Current smoker | 1 | 1 | 2
  Ex-smoker | 0 | 1 | 1
  Never smoked | 13 | 11 | 24
Educational level [Count of Participants; unit: Participants]
  Doctoral degree | 1 | 0 | 1
  Master's degree | 1 | 3 | 4
  Bachelor's degree/Junior college | 8 | 8 | 16
  Senior/Vocational high school | 4 | 1 | 5
  Junior high school | 0 | 1 | 1
Working status [Count of Participants; unit: Participants]
  Full time | 7 | 5 | 12
  Part time | 1 | 1 | 2
  Unemployed | 6 | 7 | 13
Marital status [Count of Participants; unit: Participants]
  Single | 6 | 8 | 14
  Married | 7 | 5 | 12
  Divorced | 1 | 0 | 1
Living status [Count of Participants; unit: Participants]
  Living with family | 8 | 10 | 18
  Living alone | 5 | 2 | 7
  Living in dormitory | 1 | 1 | 2
Use of laxatives [Count of Participants; unit: Participants] | 3 | 3 | 6
Menstrual cycle status [Count of Participants; unit: Participants] — Population: Only the female participant had to answer this item in the questionnaire.
  Participants
    number analyzed (Participants) | 13 | 11 | 24
    Menstruating | 10 | 7 | 17
    Peri-menopause | 1 | 3 | 4
    Post-menopause | 2 | 1 | 3
Gravidity [Count of Participants; unit: Participants] — Population: Only the female participant had to answer this item in the questionnaire.
  Participants
    number analyzed (Participants) | 13 | 11 | 24
    0 | 5 | 6 | 11
    1 | 1 | 0 | 1
    2 | 4 | 4 | 8
    3 | 1 | 0 | 1
    ≥4 | 2 | 1 | 3
Parity [Count of Participants; unit: Participants] — Population: Only the female participant had to answer this item in the questionnaire.
  Participants
    number analyzed (Participants) | 13 | 11 | 24
    0 | 5 | 6 | 11
    1 | 2 | 0 | 2
    2 | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Severity of Constipation Symptoms
Description: The Patient Assessment of Constipation Symptoms questionnaire will be used to assess the severity of constipation symptoms. This questionnaire includes a total of 12 items in 3 subscales: abdominal (4 items), rectal (3 items), and stool (5 items). Participant will be asked to rank the symptoms on a five-point Likert scale, ranging from 0 (absent) to 4 (very severe). The total score ranges from 0 to 48 which will be divided by the actual number of items answered. The higher score indicates the greater severity of constipation symptoms.
Time Frame: absolute values at 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exercise Training Group | Control Group
Number analyzed (Participants) | 14 | 13
score on a scale
  Total | 0.96 (0.59) | 0.97 (0.78)
  Abdominal | 0.63 (0.47) | 0.67 (0.98)
  Rectal | 0.67 (0.81) | 0.64 (1.17)
  Stool | 1.40 (0.94) | 1.40 (0.74)

2. Primary Outcome: Constipation Symptoms
Description: A Seven Day Bowel Diary includes items regarding the stool frequency, presence of incontinence, excessive straining, manual maneuver, or pain during defecation, and the use of laxatives.
Time Frame: absolute values at 8 weeks
Measure: Mean (Standard Deviation); unit: number/week
Arm/Group | Exercise Training Group | Control Group
Number analyzed (Participants) | 14 | 13
number/week
  Stool frequency | 5.14 (1.70) | 5.54 (1.76)
  Incontinence | 0 (0) | 0 (0)
  Excessive straining | 0.43 (0.85) | 0.62 (0.96)
  Manual maneuver | 0.07 (0.27) | 0.46 (1.66)
  Pain during defecation | 0.64 (0.93) | 0.46 (0.97)
  Use of laxatives | 1.14 (2.51) | 1.15 (2.61)

3. Primary Outcome: Constipation Symptom-Stool Consistency
Description: A Seven Day Bowel Diary includes the item regarding stool consistency. The Bristol Stool Form Scale describing the shapes and types of stools is used to evaluate stool consistency. This scale assigns a number (1-7) with 1 indicating hardest to 7 indicating loosest, to classify human feces based on its shape and and how formed or loose it is.
Time Frame: absolute values at 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exercise Training Group | Control Group
Number analyzed (Participants) | 14 | 13
score on a scale | 3.74 (1.44) | 3.46 (1.33)

4. Primary Outcome: Constipation Symptom-Time Spent During Defecation
Description: A Seven Day Bowel Diary includes items regarding time spent during defecation.
Time Frame: absolute values at 8 weeks
Measure: Mean (Standard Deviation); unit: minute/bowel movement
Arm/Group | Exercise Training Group | Control Group
Number analyzed (Participants) | 14 | 13
minute/bowel movement | 12.06 (15.15) | 9.46 (9.60)

5. Secondary Outcome: The Pelvic Floor Muscle Coordination Measured by the Pelvic Floor Muscle Coordination Scale
Description: The Pelvic Floor Muscle Coordination Scale including 5 items, respiration, pelvic floor muscle contraction, extrapelvic muscle activation, pelvic floor muscle expansion, and cough will be used to evaluate pelvic floor muscle coordination. All will be evaluated by observation. The total score ranges from 0 to 10 and a higher score indicates the poorer pelvic floor muscle coordination.
Time Frame: absolute values at 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exercise Training Group | Control Group
Number analyzed (Participants) | 14 | 13
score on a scale | 1.79 (1.25) | 2.31 (2.10)

6. Secondary Outcome: The Pelvic Floor Muscle Strength Will be Measured by Digital Rectal Examination.
Description: Resting tone, maximal voluntary contraction (MVC) of external anal sphincter and puborectalis, voluntary relaxation, and three components of defecation attempts (push effort, anal relaxation, and perineal descent) will be measured.
  Resting pressure was scored as "0=decreased", "1=normal", or "2=increased". Maximal voluntary contraction of external anal sphincter and puborectalis were scored separately for each muscle based on the International Continence Society scale criteria as "0=absent", "1=weak", "2=moderate", "3=strong". Voluntary relaxation was assessed after MVCs and scored as "0=absent", "1=partial", or "2=complete". Push effort was scored as "0=weak", "1=normal", or "2=excessive", anal relaxation was scored as "0=impaired", "1=normal", or "2=paradoxical contraction", and perineal descent was scored as "0=absent", "1=normal", or "2=excessive".
Time Frame: absolute values at 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exercise Training Group | Control Group
Number analyzed (Participants) | 14 | 13
score on a scale
  External anal sphincter resting tone | 0.71 (0.47) | 0.62 (0.51)
  Puborectalis resting tone | 1.14 (0.36) | 1.15 (0.38)
  External anal sphincter maximal voluntary contraction | 1.50 (0.65) | 1.31 (0.48)
  Puborectalis maximal voluntary contraction | 1.64 (0.50) | 1.77 (0.73)
  Voluntary relaxation | 1.71 (0.61) | 1.85 (0.38)
  Push effort | 0.86 (0.36) | 0.54 (0.52)
  Anal relaxation | 1.21 (0.43) | 1.23 (0.44)
  Perineal descent | 1.07 (0.27) | 0.85 (0.38)

7. Secondary Outcome: The Pelvic Floor Muscle Function Will be Measured Using Anorectal Manometry.
Description: Participants will be asked to relax for 10 seconds, squeeze 3 times by holding 5 seconds with 5 seconds of rest in between, and squeeze by holding the contraction for 30 seconds. Anorectal pressure will be recorded in unit of millimeter of mercury (mmHg).
Time Frame: absolute values at 8 weeks
Measure: Mean (Standard Deviation); unit: millimeter of mercury
Arm/Group | Exercise Training Group | Control Group
Number analyzed (Participants) | 14 | 13
millimeter of mercury
  Resting pressure | 2.14 (2.01) | 1.82 (1.26)
  Maximal voluntary contraction | 50.73 (40.42) | 46.52 (31.92)
  Average of maximal voluntary contraction | 23.01 (25.34) | 16.42 (17.48)

8. Secondary Outcome: The Pelvic Floor Muscle Endurance Will be Measured Using Anorectal Manometry and Stopwatch.
Description: Participants will be asked to voluntarily squeeze their pelvic floor muscles by holding the contraction for 30 seconds. Anorectal squeeze pressure is measured using an anorectal manometry. The pelvic floor muscle endurance is recorded as the time (seconds) holding at >50% of maximal voluntary contraction (squeeze pressure) in 30 seconds.
Time Frame: absolute values at 8 weeks
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Exercise Training Group | Control Group
Number analyzed (Participants) | 14 | 13
seconds | 6.78 (7.53) | 6.11 (8.04)

9. Secondary Outcome: Physical Activity Levels
Description: The International Physical Activity Questionnaire will be used to measure participants' physical activity levels. This questionnaire includes seven questions on different physical activity levels of duration and frequency and then calculated in metabolic equivalent-minutes/week. A higher score indicates a greater physical activity levels.
Time Frame: absolute values at 8 weeks
Measure: Mean (Standard Deviation); unit: metabolic equivalent-minutes/week
Arm/Group | Exercise Training Group | Control Group
Number analyzed (Participants) | 14 | 13
metabolic equivalent-minutes/week
  Total | 1069.25 (747.76) | 1253.85 (1889.07)
  Vigorous | 262.86 (354.22) | 418.46 (821.81)
  Moderate | 331.43 (275.09) | 378.46 (608.51)
  Walking | 474.96 (539.54) | 456.92 (601.91)

10. Secondary Outcome: Constipation Quality of Life
Description: Patient Assessment of Constipation Quality of Life Questionnaire will be used to evaluate the quality of life in constipation patients. This questionnaire includes a total of 28 items in 4 subscales: worries and concerns (11 items), physical discomfort (4 items), psychosocial discomfort (8 items), and satisfaction (5 items). Participants will be asked to rank how constipation affects their quality of life on a five-point Likert scale, ranging from 0 to 4. A higher score indicates greater impact on quality of life.
Time Frame: absolute values at 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exercise Training Group | Control Group
Number analyzed (Participants) | 14 | 13
score on a scale
  Total | 1.30 (0.75) | 1.60 (0.85)
  Physical discomfort | 1.16 (0.68) | 1.38 (0.88)
  Worries and concerns | 1.28 (0.97) | 1.69 (1.12)
  Satisfaction | 2.36 (0.85) | 2.71 (0.51)
  Psychosocial discomfort | 0.72 (0.70) | 0.89 (0.85)

11. Secondary Outcome: Adherence
Description: Participants in intervention group will be asked to record the number of completed home exercises (pelvic floor muscle training and walking) in the exercise diary. Adherence will be calculated separately for pelvic floor muscle training and walking as the days of home exercises completed over 56 days.
Time Frame: absolute values at 8 weeks
Population: There were three missing data of adherence (n=3) in intervention group as the participants dropped out during the eight-week program.
Measure: Count of Units; unit: days
Units Other Than Participants: days
Arm/Group | Exercise Training Group
Number analyzed (Participants) | 11
Number analyzed (days) | 56
days
  Pelvic floor muscle training | 33
  Walking | 28

ADVERSE EVENTS:
Time Frame: through 8-week program
Description: In our study, adverse events were monitored but no adverse events were reported.
Arm/Group | Exercise Training Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/13
Other Adverse Events (participants affected / at risk) | 0/14 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-25): https://cdn.clinicaltrials.gov/large-docs/02/NCT04661202/Prot_SAP_000.pdf